CLINICAL TRIAL: NCT02037191
Title: RANDOMIZED DOUBLE-BLIND STUDY MULTICENTRIQUE TESTING THE EFFICIENCY OF the METHOTREXATE AT PATIENTS AFFECTED BY GRAVE PELADE (METHOTREXATE VERSUS PLACEBO WITH SECONDARY TREATMENT BY METHOTREXATE and PREDNISONE)
Brief Title: The Efficiency Of The Methotrexate At Patients Affected By Grave Pelade
Acronym: MP3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011/121/HP
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: ALOPECIA AREATA
Keywords: ALOPECIA AREATA; TREATMENT METHOTREXATE
MeSH Terms: conditions — Alopecia Areata | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A : METHOTREXATE (Placebo Comparator): Arm A: methotrexate 20 to 25 mg / week for 6 months. Patients who will experience at least a 25% hair regrowth after the month 5 evaluation will continue methotrexate or placebo from month 6 to the end of the study (month 12).
  Non responder patients in both arms A and B will be re-randomized to receive from month 6 to the end of the study (month 12):
  * methotrexate alone or
  * methotrexate associated with prednisone 0.3 mg/Kg/day
  Interventions: Drug: Methotrexate
- ARM B : PLACEBO (Placebo Comparator): Arm B placebo Patients who will experience at least a 25% hair regrowth after the month 5 evaluation will continue methotrexate or placebo from month 6 to the end of the study (month 12).
  Non responder patients in both arms A and B will be re-randomized to receive from month 6 to the end of the study (month 12):
  * methotrexate alone or
  * methotrexate associated with prednisone 0.3 mg/Kg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Non responder patients in arm A will be re-randomized to receive from month 6 to the end of the study (month 12):
  methotrexate alone or methotrexate associated with prednisone 0.3 mg/Kg/day
  Other Names: Arm A: methotrexate 20 to 25 mg / week for 6 months.
  Arms: ARM A : METHOTREXATE
Drug: Placebo — Non responder patients in arm B will be re-randomized to receive from month 6 to the end of the study (month 12):
  methotrexate alone or methotrexate associated with prednisone 0.3 mg/Kg/day
  Arms: ARM B : PLACEBO

SUMMARY:
Alopecia areata (AA) is an auto immune disorder. Treatment of severe types remains difficult with a rate of hair regrowth which is lower than 10%. This RCT will assess the safety and efficacy of methotrexate alone or associated with low doses of prednisone versus placebo in the treatment of severe types of AA.

DETAILED DESCRIPTION:
Background: Alopecia areata (AA) is an auto immune disorder. Chronic and severe types of AA have a major impact on patients' quality of life. Treatment of severe types of AA include phototherapy, pulse IV corticosteroids, topical immunotherapy. These treatments are poorly effective in severe types of AA, since the rate of hair regrowth remains lower than 10%. Methotrexate is an immunosuppressant which is used in many autoimmune skin disorders.

Aim: To assess the safety and efficacy of methotrexate versus placebo in the treatment of severe types of AA.

Design: Patients will be randomly assigned to receive methotrexate 20 to 25 mg / week for 6 months. Patients who will experience at least a 25% hair regrowth after 5 months will continue methotrexate or placebo from month 6 to the end of the study (month 12). Non responder patients will be re randomized to receive either methotrexate alone or associated with prednisone 0.3 mg/Kg/day from month 6 to the end of the study (month 12).

Study Design Primary outcome Rate of complete or almost complete hair regrowth at the month 12 evaluation in patients treated with methotrexate or placebo who have not been re randomized after the month 5 evaluation and have staid in their initial group of randomization Secondary outcomes

1. Rate of Global Regrowth Assesment (GRA) at month 6 and 12 .
2. Delay of hair regrowth
3. Rate of relapse
4. Quality of life
5. Safety

Arm description Arm A: methotrexate 20 to 25 mg / week for 6 months. Arm B placebo Patients who will experience at least a 25% hair regrowth after the month 5 evaluation will continue methotrexate or placebo from month 6 to the end of the study (month 12).

Non responder patients in both arms A and B will be re-randomized to receive from month 6 to the end of the study (month 12):

* methotrexate alone or
* methotrexate associated with prednisone 0.3 mg/Kg/day 10 A study population Adult patients with severe types of AA evolving without hair regrowth for at least 6 months despite previous treatments with impaired quality of life

Eligibility criteria Inclusion criteria

1. age 18 TO 70 years old
2. informed consent,
3. severe type of AA defined as : 3.1 - AA totalis universalis 3.2 - evolving for more than 6 months despite previous treatments including photothérapy (PUVA oru UVB), applications of super potent topical corticosteroid ( clobetasol propionate), applications of minoxidil 5%, or IV pulse corticosteroids 3.3 - DLQI score inferior or equal to 10

Non inclusion criteria

* Pregnant or breast feeding women
* VIH + patients
* active hepatitis B or C
* treatment with immunosuppressant (ciclosporine, mycophénolate mofetil, cyclophosphamide, azathioprine, méthotrexate) within 2 months before inclusion
* severe cardiac arythma or severe cardiac insufficiency or severe coronary disease
* liver disorder
* alcool consumption
* renal failure
* Severe diabetes mellitus
* past history of severe infection
* past history of néoplasiae ( excluding BCC),
* Karnofsky index <à 50 %
* severe lung disorder
* mental impairment
* symptomatic osteoporosis
* blood cytopénia (hémoglobine < 10 g/l ; leucocytes< 3000/mm3, platelets< 100 000/mm3)
* albuminémia < 25 g/l

ELIGIBILITY:
Inclusion Criteria:

1. - age 18 to 70 years old
2. - informed consent,
3. - severe type of AA defined as : 3.1 - AA totalis universalis 3.2 - evolving for more than 6 months despite previous treatments including photothérapy (PUVA oru UVB), applications of super potent topical corticosteroid ( clobetasol propionate), applications of minoxidil 5%, or IV pulse corticosteroids 3.3 - DLQI score superior or equal to 10

Exclusion Criteria:

* Pregnant or breast feeding women
* VIH + patients
* active hepatitis B or C
* treatment with immunosuppressant (ciclosporine, mycophénolate mofetil

  , cyclophosphamide, azathioprine, méthotrexate) within 2 months before inclusion
* severe cardiac arythma or severe cardiac insufficiency or severe coronary disease
* liver disorder
* alcool consumption
* renal failure
* Severe diabetes mellitus
* past history of severe infection
* past history of néoplasiae ( excluding BCC),
* Karnofsky index <à 50 %
* severe lung disorder
* mental impairment
* symptomatic osteoporosis
* blood cytopénia (hémoglobine < 10 g/l ; leucocytes< 3000/mm3, platelets< 100 000/mm3)
* albuminémia < 25 g/l

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
OUTCOME MESURE | MONTH12
  primary outcome Rate of complete or almost complete hair regrowth at the month 12 evaluation in patients treated with methotrexate or placebo who have not been re randomized after the month 5 evaluation and have staid in their initial group of randomization

SECONDARY OUTCOMES:
SECONDARY OUTCOME MEASURE | MONTH 6 TO 12
  1 Rate of Global Regrowth Assesment (GRA) at month 6 and 12 .
  * 2 Delay of hair regrowth
  * 3 Rate of relapse
  * 4 Quality of life
  * 5 Safety

CONTACTS AND LOCATIONS:
Overall Officials: PASCAL JOLY, PROFESSOR, Principal Investigator — CHU - Hôpitaux de Rouen
Locations (2):
- France (2):
  - Head Dermatology Department, Rouen, Haute Normandie
  - CHU de Rouen - Hôpitaux de Rouen, Rouen, Seine Maritime

REFERENCES:
- [Derived] Joly P, Lafon A, Houivet E, Donnadieu N, Richard MA, Dupuy A, Delaporte E, Bernard P, Machet L, Tosti A, Del Marmol V, Grimalt R, de Viragh PA, Benichou J, Chosidow O, Assouly P, Reygagne P. Efficacy of Methotrexate Alone vs Methotrexate Plus Low-Dose Prednisone in Patients With Alopecia Areata Totalis or Universalis: A 2-Step Double-Blind Randomized Clinical Trial. JAMA Dermatol. 2023 Apr 1;159(4):403-410. doi: 10.1001/jamadermatol.2022.6687. PMID 36884234